CLINICAL TRIAL: NCT02532478
Title: Fortune of Temporary Ileostomies in Patients Treated With Laparoscopic Low Anterior Resection for Rectal Cancer
Brief Title: Fortune of Temporary Ileostomies in Patients After Rectal Cancer Surgery
Status: Completed | Type: Observational
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Nuri Okkabaz, MD, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Other Study IDs: DrLutfi
Record Dates: First submitted 2015-08-19; First posted 2015-08-25 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Loop Ileostomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Stoma reversed: Patients whose ileostomy have been closed after laparoscopic low anterior resection
- Stoma not-reversed: Patients whose ileostomy have not been closed due to some problems

SUMMARY:
The risk factors for stoma reversal failure have been rarely studied, which is probably one of the worst scenarios for a case who has a sphincter preserving procedure for a rectal cancer and is expecting to have regular bowel movements through a functional anus. Several studies have analyzed this particular issue and some have shown that up to 30% of 'temporary' stomas have never been closed. However these data have been criticized to be heterogeneous, since they have included patients with benign and malignant diseases, cases underwent elective or emergent anterior or low anterior resections or restorative proctocolectomy; and those with a colostomy or ileostomy, even an end stoma in some subjects. In addition, some studies have underlined some risk factors for the failure of stoma reversal, but they also have similar limitations as mentioned above. Finally, survival -to the best of investigators' knowledge- has never been separately studied in patients who cannot receive a stoma reversal procedure. Thus, current study aims to present a single-surgeon experience regarding the rate of diverting ileostomy takedown, the factors adversely affecting stoma reversal rate in patients underwent laparoscopic low anterior resection for rectal cancer, and accordingly to expose the fortune of these cases.

DETAILED DESCRIPTION:
Defunctioning stomas are commonly formed in order to divert the bowel stream mostly in case of distal anastomosis, particularly after a low anterior resection. It has been reported that a temporary ileostomy may decrease the risk of an anastomotic leak, which is a lethal complication. In addition, in case of an anastomotic leak, stomas may limit the septic sequence and may help the diseased anastomosis to heal or the area of inflammation to resolve. Stomas have been also shown to decrease the necessity of an urgent reoperation due to septic intra-abdominal complications that may occur after an anastomotic leak. Many believe that stoma complications are generally easily managed and reversal of stomas are associated with limited morbidity. Thus, selective or routine creation of diverting stomas have been recommended in patients underwent a low anterior resection.

The risk factors for stoma reversal failure have been rarely studied, which is probably one of the worst scenarios for a case who has a sphincter preserving procedure for a rectal cancer and is expecting to have regular bowel movements through a functional anus. Several studies have analyzed this particular issue and some have shown that up to 30% of 'temporary' stomas have never been closed. However these data have been criticized to be heterogeneous, since they have included patients with benign and malignant diseases, cases underwent elective or emergent anterior or low anterior resections or restorative proctocolectomy; and those with a colostomy or ileostomy, even an end stoma in some subjects. In addition, some studies have underlined some risk factors for the failure of stoma reversal, but they also have similar limitations as mentioned above. Finally, survival -to the best of investigators' knowledge- has never been separately studied in patients who cannot receive a stoma reversal procedure. Thus, current study aims to present a single-surgeon experience regarding the rate of diverting ileostomy takedown, the factors adversely affecting stoma reversal rate in patients underwent laparoscopic low anterior resection for rectal cancer, and accordingly to expose the fortune of these cases.

ELIGIBILITY:
Inclusion Criteria:

* All patients who received laparoscopic low anterior resection and loop ileostomy for rectal cancer, except:

Exclusion Criteria:

* patients undergoing an operation for a benign or recurrent disease or an emergent condition,
* those presenting with insitu cancer or dysplasia without an invasive cancer,
* those with cancers other than adenocarcinomas,
* those received a restorative proctocolectomy,
* those necessitated diversion for an irresectable tumor,
* those received a diverting/end colostomy or end ileostomy,
* Patients who had a recurrent disease and/or unresectable metastasis after the creation of stoma
* those received a temporary stoma during the last 12 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who underwent laparoscopic low anterior resection for rectal cancer with a diverting ileostomy between 2007 and 2014.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2007-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Stoma closure rate | up to 84 months

OTHER OUTCOMES:
Postoperative complications after primary surgery | 30 days
  not only 30-day but all in-hospital complications including readmissions
5-year overall survival | 5 years
  the time from the primary operation {laparoscopic low anterior resection} to death from any cause